CLINICAL TRIAL: NCT00031824
Title: Phase III Trial of Hydroxychloroquine + Standard Therapy for Chronic Graft-Versus-Host Disease
Brief Title: Hydroxychloroquine in Treating Patients With Newly Diagnosed Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASCT0031; COG-ASCT0031 (Other: Children's Oncology Group); CCG-S9701 (Other: Children's Cancer Group); NCI-P02-0213
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclosporine; Hydroxychloroquine; Prednisone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclosporine
Drug: hydroxychloroquine
Drug: prednisone
Drug: tacrolimus

SUMMARY:
RATIONALE: Hydroxychloroquine may decrease the immune response and be effective in treating chronic graft-versus-host disease. It is not yet known if standard therapy for graft-versus-host disease is more effective with or without hydroxychloroquine.

PURPOSE: Randomized phase III trial to compare the effectiveness of standard therapy alone with that of standard therapy plus hydroxychloroquine in treating patients who have newly diagnosed chronic graft-versus-host disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of prednisone and cyclosporine with vs without hydroxychloroquine in patients with newly diagnosed extensive chronic graft-versus-host disease (GVHD).

Secondary

* Compare the event-free and overall survival in patients treated with these regimens.
* Compare the health-related quality of life, including longitudinal change in and magnitude of persistent disability, in patients treated with these regimens.
* Correlate cytokine levels and T-helper cell subtypes with chronic GVHD activity and response in patients treated with these regimens.
* Correlate whole blood hydroxychloroquine levels with response and toxicity in patients treated with these regimens.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are randomized to one of two treatment arms.

Patients may receive standard therapy comprising prednisone orally or IV 2-3 times daily or every other day and cyclosporine orally or IV twice daily or tacrolimus orally twice daily or IV by continuous infusion before randomization. Patients not receiving cyclosporine or tacrolimus prior to randomization may receive cyclosporine or tacrolimus after randomization according to institutional preference.

* Arm I: Within 10-14 days of beginning therapy with prednisone and cyclosporine or tacrolimus, patients receive oral hydroxychloroquine twice daily.
* Arm II: Patients receive standard therapy with prednisone and cyclosporine or tacrolimus as in arm I and oral placebo twice daily.

In both arms, treatment continues for 9 months in the absence of disease progression or unacceptable toxicity. Patients with no response after 2 months of therapy are taken off study.

Quality of life is assessed at baseline, 1 month, 9 months, and 1 year.

Patients are followed every month for 3 months and at 9 months.

PROJECTED ACCRUAL: A total of 232 patients (116 per treatment arm) will be accrued for this study within 3.6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* newly diagnosed extensive chronic graft-versus-host disease (GVHD) of ≥ 1 organ system (e.g., lip, skin, or liver) documented by all of the following:

  * Clinicopathologic features of GVHD, including involvement of any of the following organ systems:

    * Skin changes
    * Oral changes
    * Hepatic involvement
    * Gastrointestinal involvement
    * Sicca syndrome
    * Pulmonary involvement
    * Myofascial
    * Skeletal
    * Other inflammatory conditions (e.g., myositis, arthritis, polyserositis, or unexplained pericardial, pleural, or peritoneal effusions)
    * Autoantibodies
  * Extent of disease, defined according to the following classification:

    * Limited chronic GVHD, defined by 1 of the following:

      * Localized skin involvement and/or liver dysfunction
      * Involvement of only 1 target organ
    * Extensive chronic GVHD, defined by 1 of the following:

      * Generalized skin involvement of ≥ 50% of body surface area
      * Localized skin involvement and/or liver dysfunction AND ≥ 1 of the following:

        * Liver histology showing chronic aggressive hepatitis, bridging necrosis, or cirrhosis
        * Eye involvement (Schirmer's test with < 5 mm wetting)
        * Involvement of minor salivary glands or oral mucosa on lip biopsy
        * Involvement of any other target organs
      * Involvement of ≥ 2 target organs
  * Timing of onset, including onset of any of the following types:

    * Progressive onset defined as, evolving directly from acute GVHD, commonly with the development of typical manifestations such as oral or skin lichenoid changes or sclerodermatous skin changes
    * Quiescent onset, defined as developing after the resolution of acute GVHD
    * De novo onset, defined as developing with no prior history of acute GVHD
* Must have ≥ 1 typical clinical manifestation of chronic GVHD that differs from that of acute GVHD (e.g., rash, anorexia, nausea, emesis, diarrhea, abdominal pain, or cholestasis)

  * Symptoms of acute GVHD allowed at the time of diagnosis of chronic GVHD
* Prior allogeneic bone marrow, peripheral blood stem cell, or cord blood transplantation from a family member or unrelated donor for malignancy required NOTE: *Histologic confirmation may be "consistent with GVHD"

PATIENT CHARACTERISTICS:

Age:

* 1 to 29

Performance status:

* Lansky 50-100% OR
* Karnofsky 50-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count ≥ 1,000/mm^3, unless due to chronic GVHD (i.e., autoimmune neutropenia or bone marrow suppression)

Hepatic:

* See Disease Characteristics

Renal:

* Creatinine < 1.5 times upper limit of normal OR
* Creatinine clearance ≥ 60 mL/min

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No lysosomal storage disorder
* No uncontrolled infection (e.g., persistent bacterial, fungal, or viral infection despite appropriate antimicrobial therapy)
* No G6PD deficiency
* No history of psoriasis or porphyria
* No hypersensitivity to 4-aminoquinolines
* No prior retinal or visual field changes due to 4-aminoquinolines

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent daclizumab or infliximab
* No concurrent thalidomide

Chemotherapy:

* Not specified

Endocrine therapy:

* Prior topical steroids for treatment of extensive chronic GVHD allowed
* Prior adjustment to prednisone dose allowed if done as a reversal of a taper
* Prior steroids (prednisone ≤ 1 mg/kg/day (or equivalent) for symptom management for up to 1 week before study entry allowed
* Concurrent steroids for treatment and/or prophylaxis of acute GVHD allowed if prednisone dose is ≤ 2 mg/kg/day (or equivalent)
* Concurrent topical steroids allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior treatment for extensive chronic GVHD except the following:

  * Topical treatment (e.g., tacrolimus ointment or pimecrolimus cream)
  * Adjustments of cyclosporine or tacrolimus doses for GVHD prophylaxis or treatment of acute GVHD
* Concurrent cyclosporine or tacrolimus allowed

  * Cyclosporine must have been started before study entry
* No other concurrent systemic or topical immunosuppressants, including any of the following:

  * Azathioprine
  * Mycophenolate mofetil
  * Psoralen-ultraviolet light therapy
  * Photopheresis
* No administration of any of the following for 1 hour before until 2 hours after study drug administration:

  * Antacids
  * Sucralfate
  * Cholestyramine
  * Bicarbonate

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2002-04; Primary Completion 2005-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Length of study

SECONDARY OUTCOMES:
Compare the efficacy of a two-drug regimen | Length of study
  Compare the efficacy of a two-drug regimen including prednisone and cyclosporine versus that of a three-drug regimen including hydroxychloroquine, prednisone, and cyclosporine in patients treated for newly-diagnosed extensive chronic GVHD.
Compare conventional outcomes measures | Length of study
  Compare conventional outcomes measures (event-free survival, overall survival) and health-related quality-of-life (HRQL), including longitudinal change in and magnitude of persistent disability, for the two-drug versus the three-drug regimen.
To determine if cytokine levels and T helper cell subtypes (Th1 and Th2) correlate with chronic GVHD activity and response | Length of study
Determine if whole blood hydroxychloroquine levels correlate with response and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L. Gilman, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (104):
- United States (89):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University Medical Center at Princeton, Los Angeles, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Presbyterian - St. Luke's Medical Center, Colorado Springs, Colorado
  - Children's Hospital Cancer Center, Denver, Colorado
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics - Minneapolis/St. Paul, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Children's Hospital at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Pediatric Hematology and Oncology Associates of South Texas, PLLC, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- Starship Children's Health, Auckland, New Zealand
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Gilman AL, Schultz KR, Goldman FD, Sale GE, Krailo MD, Chen Z, Langholz B, Jacobsohn DA, Chan KW, Ryan RE, Kellick M, Neudorf SM, Godder K, Sandler ES, Sahdev I, Grupp SA, Sanders JE, Wall DA. Randomized trial of hydroxychloroquine for newly diagnosed chronic graft-versus-host disease in children: a Children's Oncology Group study. Biol Blood Marrow Transplant. 2012 Jan;18(1):84-91. doi: 10.1016/j.bbmt.2011.05.016. Epub 2011 May 30. PMID 21689773
- [Result] Rozmus J, Schultz KR, Wynne K, Kariminia A, Satyanarayana P, Krailo M, Grupp SA, Gilman AL, Goldman FD. Early and late extensive chronic graft-versus-host disease in children is characterized by different Th1/Th2 cytokine profiles: findings of the Children's Oncology Group Study ASCT0031. Biol Blood Marrow Transplant. 2011 Dec;17(12):1804-13. doi: 10.1016/j.bbmt.2011.05.011. Epub 2011 May 25. PMID 21669298
- [Result] Hall MJ, Reid JE, Wenstrup RJ. Prevalence of BRCA1 and BRCA2 mutations in women with breast carcinoma In Situ and referred for genetic testing. Cancer Prev Res (Phila). 2010 Dec;3(12):1579-85. doi: 10.1158/1940-6207.CAPR-09-0218. PMID 21149333
- [Result] Fujii H, Cuvelier G, She K, Aslanian S, Shimizu H, Kariminia A, Krailo M, Chen Z, McMaster R, Bergman A, Goldman F, Grupp SA, Wall DA, Gilman AL, Schultz KR. Biomarkers in newly diagnosed pediatric-extensive chronic graft-versus-host disease: a report from the Children's Oncology Group. Blood. 2008 Mar 15;111(6):3276-85. doi: 10.1182/blood-2007-08-106286. Epub 2007 Oct 9. PMID 17925486